CLINICAL TRIAL: NCT05788965
Title: Efficacy and Safety of GLP-1 Agonist Therapy in Overweight and Obese Subjects With Cystic Fibrosis-related Diabetes: a Pilot Study
Brief Title: Semaglutide in CFRD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MED-2023-29616
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis-related Diabetes
Keywords: CFRD
MeSH Terms: conditions — Cystic Fibrosis | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: This open label, single arm pilot study, will examine the safety and tolerability of GLP-1RA semaglutide as an add-on therapy to insulin for overweight/obese adult patients with CFRD.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): Semaglutide 1 mg once weekly subcutaneous injection
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — glucagon-like peptide 1 (GLP-1) receptor agonist
  Other Names: GLP-1 RA; Semaglutide Injectable Product

SUMMARY:
This open label, single arm pilot study, will examine the safety and tolerability of GLP-1RA semaglutide as an add-on therapy to insulin for overweight/obese adult patients with cystic fibrosis related diabetes (CFRD).

DETAILED DESCRIPTION:
The overall goal of this proposal is to collect pilot data for safety and feasibility metrics to support a future larger randomized controlled trial. In this study, we will examine the safety and tolerability of GLP-1RA semaglutide as an add-on therapy to insulin for overweight/obese adult patients with CFRD. We hypothesize that weekly administration of the long-acting GLP-1RA semaglutide to overweight/obese CFRD patients will be safe and well tolerated.

Specific Aim 1: Collect pilot data on the safety and feasibility of weekly semaglutide therapy in overweight and obese patients with CFRD to support a future larger randomized controlled trial.

Hypothesis 1: Weekly therapy with GLP-1RA semaglutide will be safe and well tolerated in overweight/obese adults with CFRD.

Specific Aim 2: Collect preliminary data to examine the impact of semaglutide therapy on insulin secretion, glucagon and glucose levels as measured by oral glucose tolerance test (OGTT), and on glycemic outcomes as measured by continuous glucose monitoring (CGM) and HbA1c.

Hypothesis 2a: Treatment with semaglutide will lower glucose levels, and increase insulin and C-peptide area under the curve (AUC) during the OGTT as compared to baseline.

Hypothesis 2b: Treatment with semaglutide will improve glycemic control as indicated by time in range on CGM and HbA1c

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18 years or older with CFRD and on insulin treatment
* BMI >26 kg/m2
* Diagnosis of pancreatic insufficiency (based on treatment with pancreatic enzyme replacement therapy)
* A participant who is capable of becoming pregnant must agree to take precautions that are effective in preventing pregnancy throughout this study. These methods could include one of the following 1. Complete abstinence from sexual intercourse; 2. Oral, injectable, or implanted hormonal contraceptives 3. Intrauterine device 4. Tubal ligation

Exclusion Criteria:

* personal or family history of medullary thyroid cancer or multiple endocrine neoplasia syndrome type 2 (MEN2)
* acute pulmonary exacerbation requiring IV antibiotics or systemic glucocorticoids within 4 weeks prior to baseline study procedures
* gastrointestinal(GI) symptom exacerbation defined by current nausea/vomiting or diarrhea at the baseline assessment
* history of chronic GI problems requiring hospitalization in the 1 year prior to baseline
* history of clinically symptomatic pancreatitis
* history of clinically significant gastroparesis
* history of eating disorders
* less than 24 weeks since start of a new CFTR corrector/modulator therapy
* pregnancy or lactation
* severe CF liver disease
* chronic kidney disease
* history of suicide attempts or active suicidal ideation
* Non-English speakers and those unable to read in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Moheet, MBBS, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

RESULTS

PARTICIPANT FLOW:
Groups:
- Semaglutide Treatment: This open label, single arm pilot study, will examine the safety and tolerability of GLP-1RA semaglutide as an add-on therapy to insulin for overweight/obese adult patients with CFRD.
  Semaglutide: glucagon-like peptide 1 (GLP-1) receptor agonist
Period: Overall Study
Arm/Group | Semaglutide Treatment
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Semaglutide Treatment
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Change in weight before and 12 weeks post treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Semaglutide Treatment
Number analyzed (Participants) | 8
kilograms | -4.6 (1.9)

2. Primary Outcome: BMI (kg/m2)
Description: Change in BMI before and 12 weeks post treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Semaglutide Treatment
Number analyzed (Participants) | 8
kg/m2 | -1.8 (0.9)

3. Secondary Outcome: CGM % Time in Target TIR)
Description: Change in CGM TIR before and 12 weeks post treatment. Outcome reflects the change in continuous glucose monitoring (CGM) time in range (TIR), measured at baseline and again 12 weeks after treatment initiation.
  TIR is defined as the percentage of time glucose values are between 70 and 180 mg/dL
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage time in target
Arm/Group | Semaglutide Treatment
Number analyzed (Participants) | 8
percentage time in target | 7 (10.5)

4. Secondary Outcome: A1c
Description: change in the percent of HbA1c before and 12 weeks post treatment
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: change in the percent of HbA1c
Arm/Group | Semaglutide Treatment
Number analyzed (Participants) | 8
change in the percent of HbA1c | -0.3 (0.3)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Semaglutide Treatment
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide Treatment (N=8)
Nausea (Gastrointestinal disorders) | 5 (8)
Constipation (Gastrointestinal disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Heartburn (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
there was no placebo control

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT05788965/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-13): https://cdn.clinicaltrials.gov/large-docs/65/NCT05788965/ICF_001.pdf